CLINICAL TRIAL: NCT04034160
Title: A Comparison of the Rise of Serum Lipids, Glucose, and Hs-CRP Levels After Consumption of a Beef Burger Versus a Vegetarian Burger
Brief Title: Beef Burger Versus a Vegetarian Burger
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Cindy Kosch, Chair and Program Director, Department of Nutrition and Dietetics, School of Allied Health Professionals, Loma Linda University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 5190215
Record Dates: First submitted 2019-07-19; First posted 2019-07-26 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- burger consumption group (Experimental): Each participant will consume a burger with a whole wheat bun, lettuce, tomatoes, and vegan mayonnaise (free of cholesterol) for one meal. The burger patty will be 4 ounces. The beef patty (Beef Patty Chuck) will be 80% lean and 20% fat.
  Interventions: Other: vegetarian burger
- vegetarian burger consumption group (Active Comparator): Each participant will consume a burger with a whole wheat bun, lettuce, tomatoes, and vegan mayonnaise (free of cholesterol) for one meal. The burger patty will be 4 ounces. The vegetarian patty (Impossible Burger) will be 18% fat.
  Interventions: Other: beef burger

INTERVENTIONS:
Other: vegetarian burger — A finger prick test will be used to determine baseline levels measurements for serum lipids, glucose, and hs-CRP levels. Group 1 will be given vegetarian burgers to consume. Participants will need to remain in the room for 2 hours, postprandial (they may study, watch a movie, etc). They will not be allowed to consume anything except for water during this time. After consumption of burger, at 30 min, 60 min, 120 min, finger prick tests will be used to obtain blood. Participants will also be asked to try and identify the burger they consumed and rate the taste of the burger. Visit 2 will take approximately 3 hours.
  * Participants will be directed to fast for 8 hours prior to Visit 3 (the following week).
  * Visit 3: We will repeat the same procedure as Visit 2. However, this time the burgers will be switched.
  Arms: burger consumption group
Other: beef burger — A finger prick test will be used to determine baseline levels measurements for serum lipids, glucose, and hs-CRP levels. Group 2 will be given beef burgers to consume. Participants will need to remain in the room for 2 hours, postprandial (they may study, watch a movie, etc). They will not be allowed to consume anything except for water during this time. After consumption of burger, at 30 min, 60 min, 120 min, finger prick tests will be used to obtain blood. Participants will also be asked to try and identify the burger they consumed and rate the taste of the burger. Visit 2 will take approximately 3 hours.
  * Participants will be directed to fast for 8 hours prior to Visit 3 (the following week).
  * Visit 3: We will repeat the same procedure as Visit 2. However, this time the burgers will be switched.
  Arms: vegetarian burger consumption group

SUMMARY:
The purpose of this graduate student research study is to compare the rise of serum lipids, glucose, and hs-CRP levels after consumption of a beef burger versus a vegetarian burger in healthy adults between the ages of 21 and 55

DETAILED DESCRIPTION:
Visit 1

* Sign an informed consent.
* Complete a brief questionnaire about demographics (age, gender, and race), eating habits, physical activity level, and medical history (known allergies, and history of dyslipidemia, diabetes mellitus, or arthritis)
* Will be directed to fast for 8 hours prior to Visit 2. Visit 2
* Be randomized into either Group 1 or Group 2. One group will eat the beef burger first and the other group will eat the vegetarian burger first.
* Fill out a questionnaire on number of hours slept and current stress level.
* Take a finger prick test (tiny drop of blood) to determine baseline measurements for serum lipids, glucose, and hs-CRP levels.
* Consume either a beef burger or vegetarian burger.
* Afterwards, remain in Nichol Hall, Room A112, for 2 hours (may study, watch a movie, etc.).
* May not consume anything except for water.
* After 30 min, 60 min, 120 min, finger prick tests will be used to measure post-consumption serum lipids, glucose, and hs-CRP levels.
* Will be asked to try and identify burger consumed and rate the taste of the burger.
* Will be directed to fast for 8 hours prior to Visit 3. Visit 3
* Repeat the same procedure as Visit 2. However, this time the burgers will be switched.

ELIGIBILITY:
Inclusion criteria:

* Healthy adults between 21 and 55 years of age
* Consume both beef and vegetarian products
* No distaste for whole wheat buns, lettuce, soy, tomatoes, or vegan mayonnaise
* Willing to abstain from caffeine and exercise the morning of visits (2 days)

Exclusion criteria:

* Those allergic to the following food items:

  * Gluten
  * Lettuce
  * Soy
  * Tomatoes
  * Vegan Mayonnaise
* Have a known history of dyslipidemia, diabetes mellitus, or arthritis

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-01-28 (Actual); Study Completion 2020-01-28 (Actual)

PRIMARY OUTCOMES:
serum lipid panel concentration | change between visit 2(up to 7 days after initial study enrollment) and visit 3(exactly 7 days after Visit 2)
  Finger prick tests (tiny drop of blood) will be used to measure serum lipids at baseline, and then at 30 minutes, 60 minutes, and 120 minutes postprandial to determine each participant's lipid profile.

SECONDARY OUTCOMES:
glucose blood concentration | change between visit 2(up to 7 days after initial study enrollment) and visit 3(exactly 7 days after Visit 2)
  Finger prick tests (tiny drop of blood) will be used to measure glucose at baseline, and then at 30 minutes, 60 minutes, and 120 minutes postprandial to determine each participant's lipid profile.
hs-CRP blood concentration | change between visit 2(up to 7 days after initial study enrollment) and visit 3(exactly 7 days after Visit 2)
  Finger prick tests (tiny drop of blood) will be used to measure hs-CRP at baseline, and then at 30 minutes, 60 minutes, and 120 minutes postprandial to determine each participant's lipid profile.

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Kosch, MS, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States